CLINICAL TRIAL: NCT06530069
Title: Exploring the Risk Factors of Otomycosis: A Case-Control Study
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: xmzsyyky-2024-078
Record Dates: First submitted 2024-05-30; First posted 2024-07-31 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Otomycosis
Keywords: Otomycosis; predisposing factor
MeSH Terms: conditions — Otomycosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: this group consists of patients who have been diagnosed with otomycosis.Observational exposures: Ear cleaning, swimming, wearing earphones, diabetes, immunosuppression, antibiotic ear drops, narrowing of the external auditory canal, etc.
  Interventions: Other: exposures
- Control Group: This group includes healthy individuals who have not been diagnosed with otomycosis during medical examinations.Observational exposures: Ear cleaning, swimming, wearing earphones, diabetes, immunosuppression, antibiotic ear drops, narrowing of the external auditory canal, etc.
  Interventions: Other: exposures

INTERVENTIONS:
Other: exposures — exposures: Ear cleaning, swimming, wearing earphones, diabetes, immunosuppression, antibiotic ear drops, narrowing of the external auditory canal, etc.

SUMMARY:
The goal of this observational study is to explore the risk factors of fungal otitis externa in the fungal otitis externa patients The main question it aims to answer is:

What behaviors lead to the occurrence of fungal otitis externa? Participants will complete a detailed questionnaire survey. If there is a comparison group: Researchers will compare the healthy group and the disease group to see if there are any differences.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms in the case group include tinnitus, ear fullness or blockage, itching, ear pain, discharge, and hearing loss. Physical examination reveals the presence of hyphae, scabs, secretions, masses, pus, red skin, erosion, swelling, or granulation in the ear canal. Laboratory fungal cultures must be positive. The control group does not have the aforementioned ear symptoms and has not sought medical attention for ear-related symptoms.

Exclusion Criteria:

* Patients with otitis media, tympanic membrane perforation, or post-radiotherapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our institution is a tertiary first-class comprehensive hospital. Both the disease group and the control group are seen and screened at our facility
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Odds Ratio | 1month
  The ratio of exposed to non-exposed individuals in the case group divided by the ratio of exposed to non-exposed individuals in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Chunsheng Ye, MD, Principal Investigator — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital of Xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available within six months after the completion of the study and will remain accessible for at least ten years.
Access Criteria: The data will be open to peer-reviewed researchers. Researchers requesting access to the data must submit a research proposal and pass our review process. All data requestors must also adhere to a data use agreement.
URL: http://www.medresman.org